CLINICAL TRIAL: NCT04611815
Title: Does Robotic-assisted Total Knee Arthroplasty Improves Functional Outcome and Gait Pattern in Comparison to Conventional Total Knee Arthroplasty With Use of Bicruciate-stabilized (BS) Implant? Randmized-controlled Trial
Brief Title: Robotic-assisted Total Knee Arthroplasty vs. Conventional One
Acronym: RATKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WarsawMU/RATKA
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Osteo Arthritis Knee; Knee Arthritis; Knee Pain Chronic
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant will not be informed whether theis surgery was performed with robotics assist.
  Outcomes Assessor, Care provider, Investigator will not be informed which type of prosthesis was used in particular patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic-assisted total knee arthroplasty (Active Comparator): Patients undergoing robotic-assisted total knee arthroplasty with use of Journey II BCS implants
  Interventions: Procedure: Total knee arthroplasty; Diagnostic Test: Computer tomography scan; Diagnostic Test: biomechanical assesment
- Conventional total knee arthroplasty (Active Comparator): Patients undergoing conventional total knee arthroplasty with use of Journey II BCS implants
  Interventions: Procedure: Total knee arthroplasty; Diagnostic Test: Computer tomography scan; Diagnostic Test: biomechanical assesment

INTERVENTIONS:
Procedure: Total knee arthroplasty — Participant will undergo robotic-assisted or conventional total knee arthroplasty
Diagnostic Test: Computer tomography scan — CT scans of the affected knee joint before and after the surgical procedure
Diagnostic Test: biomechanical assesment — Participants will be asked to perform biomechanical assesment before and following surgery at baseline, 6-8 weeks and 6-months postoperatively

SUMMARY:
This study compares and evaluates differences in movement analysis, patient-reported outcome and radiological assesment between patients undergoing robotic-assisted total knee arthroplasty and conventional one.

DETAILED DESCRIPTION:
Osteoarthritis causes the joints to become painful and stiff. Osteoarthritis of the knee is a common condition that is expected to be a lot more frequent in the next two decades. As a consequence, an increase of total knee replacement surgery is predicted. Total knee replacement surgery is offered when knee pain and stiffness caused by osteoarthritis can no longer be managed and these symptoms significantly impact on an individual's normal activities of daily living. Most total knee replacements are successful but up to 34% of all patients have poor functional outcomes following surgery. This leaves affected people at a greater risk of reduced physical activity and thus impacts longer-term general health. Poor outcomes are therefore of importance to patients and have a considerable financial and service-provision impact on National Health Service (NHS) care. While patient-related characteristics and their relationship to patient outcomes have been identified, few studies have been undertaken to determine how kinematic outcomes (how the prosthetic knee moves) are related to functional outcome and patient satisfaction. The kinematic outcome of a total knee replacement is hypothesised to relate to both the structural design (shape) of the implant and the surgical procedure itself. In recent years, there has been development of high technology tools to help surgeon restoring proper joint biomechanics. Nowadays on the market there are several robots designed to fulfill this function. To date, no studies have investigated the kinematic outcomes of robotic-assisted total knee arthroplasty in comparison to conventional surgery. Whilst it is known that long term success of total knee replacement depends largely upon correct alignment of the prosthesis components during surgery, no studies have looked at the anatomical alignments of the osteoarthritic knee prior to undergoing surgery (using Computerised Tomography (CT) scanning). The aim of the study is to examine relationships between movement analysis (kinematic and functional outcomes), patient reported outcome measures (PROMS) with use of the combination of either Oxford score or KOOS score with addition of WOMAC and Lysholm scores and CT measurement, both pre- and post-operatively, between robotic-assisted total knee arthroplasty and conventional surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Listed for a primary total knee replacement (TKR)
2. Indication for the TKR is primary osteoarthritis of the knee joint involving one or more compartments
3. Aged 18 or over
4. Patient willing to provide full informed consent to the trial

Exclusion Criteria:

1. Listed for a single-stage one-sided TKR procedure
2. Severe symptoms in the contralateral knee so as to require staged bilateral knee replacements within 6 months of the primary procedure
3. Fixed flexion deformity of 15 degrees or greater who will require excessive resection of the distal femur
4. Clinically assessed uncorrectable varus/valgus deformity of 15 degrees or greater
5. Any co-morbidity which, in the opinion of the investigator, is severe enough to present an unacceptable risk to the patient's safety
6. Inflammatory arthritis
7. Previous septic arthritis in the affected knee joint
8. Previous surgery to the collateral ligaments of the affected knee
9. A contralateral total knee replacement that has been implanted less than one year from the date of consultation
10. A contralateral total knee replacement that is severely painful
11. Patients on warfarin or novel oral anticoagulants (NOACs)
12. Will not be resident in the catchment area for at least 6 months post-surgery
13. Undertaking the surgery as a private patient
14. Patients who, in the opinion of the clinical staff, do not have capacity to consent
15. Patients who are pregnant
16. Unable to understand written and spoken Polish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in patients reported outcome measures - Oxford Knee Score (OKS) | At baseline (preoperatively), 6-8 weeks and 12 months postoperatively.
  To explore differences between outcome in patients treated with RATKA and conventional total knee arthroplasty. Results range from 0 to 48, with higher scores corresponding to better outcomes.
Changes in patients reported outcome measures - Knee injury and Osteoarthritis Outcome Score (KOOS) | At baseline, 6-8 weeks post-operatively and 12 months post-operatively.
  To explore differences between outcome in patients treated with RATKA and conventional total knee arthroplasty. Results range from 0 to 100, with higher scores corresponding to better outcomes.
Changes in patients reported outcome measures - Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | At baseline, 6-8 weeks post-operatively and 12 months post-operatively.
  To explore differences between outcome in patients treated with RATKA and conventional total knee arthroplasty. Results range from 0 to 96, with lower scores corresponding to better outcomes.
Changes in patients reported outcome measures - Lysholm knee scoring scale | At baseline, 6-8 weeks post-operatively and 12 months post-operatively.
  To explore differences between outcome in patients treated with RATKA and conventional total knee arthroplasty. Results range from 0 to 100, with higher scores corresponding to better outcomes.
Changes in patients range of motion (ROM) | At baseline, 6-8 weeks post-operatively and 12 months post-operatively.
  To explore differences between outcome in patients treated with RATKA and conventional total knee arthroplasty. Results range from 0 to 100, with higher scores corresponding to better outcomes.
*We take into consideration the possible use of other PROM questionnaires and analysis of different adverse events depending on the unpredictable circumstances. | At baseline, 6-8 weeks post-operatively and 12 months post-operatively.
  To explore differences between outcome in patients treated with RATKA and conventional total knee arthroplasty. Results range from 0 to 100, with higher scores corresponding to better outcomes.

SECONDARY OUTCOMES:
Changes in patients reported outcome measures - Oxford Knee Score (OKS) | [Time Frame: 1 week and 6-8 weeks post-operatively]
  To explore differences between outcome in patients treated with RATKA and conventional total knee arthroplasty. Results range from 0 to 48, with higher scores corresponding to better outcomes.
Changes in patients reported outcomes - Oxford Knee Score Activity & Participation Questionnaire (OKS_APQ) | Time Frame: 1 week, 6-8 weeks and 6 months post- operatively
  To explore differences in higher levels of activity and social participation
Changes in patients reported outcomes - Forgotten Joint Score (FJS) | Time Frame: 6-8 weeks and 6 months post-operatively
  To explore differences in patient's ability to forget about a joint as a result of successful treatment. Results range from 0 to 100, with higher scores corresponding to better outcomes.
Changes in patients reported outcomes - UCLA (University of California) score | Time Frame: 6-8 weeks and 12 months post-operatively
  To explore differences in patient's physical activity. Results range from 0 to 10, with higher scores corresponding to better outcomes.
Changes in knee range of motion | Time Frame: preoperatively, 6-8 weeks and 12 months post-operatively
  To explore differences in range of motion (flexion and extension)
Changes in pain medication | Time Frame: 1 week, 6-8 weeks and 3-6 months post-operatively
  To asses evolution of post-operative knee pain
arthroplasty related complications | Time Frame: 1 week post- operatively, 6-8 weeks post-operatively and 6-12 months post-operatively
  To count and asses all complications that may occur during surgery and in postoperative period
arthroplasty revision surgeries | Time Frame: 1 week, 6-8 weeks and 12 months post-operatively
  To count and asses the reason of all revision surgeries that may occur during postoperative period
walking abilities | Time Frame: 6-8 weeks and 12 months post-operatively
  To asses "up and go" time
Length of hospital stay | Time Frame: from baseline to discharge from hospital ranging averagely from 1 up to 7 days postoperatively
  To measure number of days counting from surgery to the discharge
Biomechanical 3D motion and emg walking outcomes | Time Frame: at baseline, 6-8 weeks and 12 months post-operatively
  Overground walking is measured using 3D Motion analysis and electromyography (EMG)
Radiological outcome on CT scans | Time Frame: at baseline preoperatively and 6 weeks post- operatively
  Rotational alignment of the total knee component is assessed by measuring the femoral antetorsion, Alignment of the total knee component is assessed by measuring the tibial tubercle-trochlear groove distance (TT-TG)
6- minute walking abilities | Time Frame: 6-8 weeks and 12 months post-operatively
  to asses pace and model of 6-minute walk
Biomechanical stair climbing outcomes | Time Frame: at baseline, 6-8 weeks and 12 months post-operatively
  Stair climbing and descending is measured using 3D Motion analysis and EMG
Biomechanical static balance outcomes | Time Frame: at baseline, 6-8 weeks and 12 months post-operatively
  Static balance is measured using a force plate
Biomechanical dynamic balance outcomes | Time Frame: at baseline, 6-8 weeks and 12 months post-operatively
  Dynamic balance is measured using a force plate and the modified Star Excursion Balance Test (mSEBT)
Leg muscle strength outcomes | Time Frame: at baseline, 6-8 weeks and 12 months post-operatively
  Leg muscle strength measured using maximal voluntary isometric contraction (MVIC) test of the hamstring and quadriceps muscles on both limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz M. Maciąg, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided